CLINICAL TRIAL: NCT00046215
Title: Effect of Transcranial Magnetic Stimulation to Dorsal Premotor Cortex on Motor Imagination
Brief Title: Transcranial Magnetic Stimulation to Study Imagination of Movement
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 020312; 02-N-0312
Record Dates: First submitted 2002-09-21; First posted 2002-09-23 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2003-11

CONDITIONS: Healthy
Keywords: Virtual Lesion Study; Motor Imagery; Primary Motor Cortex; Motor Inhibition; Motor Execution; Healthy Volunteer

SUMMARY:
This study will use transcranial magnetic stimulation (TMS) to examine the relationship between cognitive processing and motor control by determining whether a part of the brain called the premotor cortex is essential to imagining movement. TMS, described below, is a method of brain stimulation that can temporarily inhibit brain functions of the area underlying the stimulator.

Healthy right-handed normal volunteers may be eligible for this study. Candidates will be screened with a medical history, neurological examination, and test of finger dexterity.

Participants will perform a sequential finger tapping movement in response to a series of numbers (stimuli) displayed on a computer monitor. After 10 stimuli, they will be asked which finger they tapped last. They will then imagine the same finger tapping movement and will be asked which finger they tapped last in their imagination. During these exercises, participants will undergo transcranial magnetic stimulation. For this procedure, the subject is seated comfortably in a chair. A wire coil is placed on the scalp and a brief electrical current is passed through the coil, creating a magnetic pulse that passes into the brain. This generates a very small electrical current in the brain, which briefly disrupts the function of the brain cells in the stimulated area. The stimulation may cause twitching in arm or leg muscles. During the stimulation, the electrical activity of muscles is recorded with a computer or other recording device, using electrodes attached to the skin with tape.

Subjects will complete eight experimental blocks of testing. One block consists of 20 experimental trials, with each trial lasting about 10 seconds. Five pairs of TMS stimuli are given per trial, with pulses delivered in short bursts of one second each. After each block, subjects draw a mark on a line on paper, showing how much attention they are paying, how much fatigue they are experiencing, and how well they think they are executing the tasks. Each TMS session takes up to 3.5 hours.

Before the TMS session, participants will undergo magnetic resonance imaging (MRI) for use in determining proper placement of the TMS coil. MRI uses a strong magnetic field and radio waves to obtain images of body organs and tissues. For this procedure, the subject lies still in a narrow metal cylinder (the scanner) for about 30 minutes during the scan.

DETAILED DESCRIPTION:
A high-level of motor control often requires complex processing of sensory information, which likely corresponds to the neural correlates for mental imagery of movement. Such cognitive aspects of motor control may underlie other cognitive functions, such as mental calculation. The present transcranial magnetic stimulation (TMS) study is aimed to characterize the relation between cognitive processing and motor control. Based on our previous results from neuroimaging experiments, we hypothesize that the ability to process information for motor imagery would primarily be associated with the dorsal lateral premotor context (PMd) as well as the posterior parietal cortex. TMS will be used to disrupt neural processes in the limited brain structures under the coil for a short period of time (virtual lesion study). For this proposal, 15 healthy subjects will perform number-guided motor execution/imagery tasks. Both tasks will be guided by 10 visual number stimuli presented at a rate of 1.0 Hz. For the test TMS stimuli, a paired TMS stimulation will be delivered to either M1 or PMd100 (to) 150 milliseconds after 5 of the visual number stimuli. The frequency of TMS stimulation will be 1.0 Hz on average for a short period of time (10 seconds). Measurement will be accuracy of the task performance under the TMS stimulation as compared with a sham condition. We expect that the TMS stimulation to PMd will interfere with the performance of motor imagery more than the performance of motor execution. The present study will clarify the neural correlates underlying the ability of imagining movement, which is now drawing growing attention in the neuroscience community.

ELIGIBILITY:
INCLUSION CRITERIA:

We will only recruit right-handed subjects as assessed by Edinburgh handedness inventory (Oldfield, 1971). We will also administer a simple version of the tapping task and assess their dexterity to select subjects consistent with the digit skills required.

EXCLUSION CRITERIA:

Contraindications for TMS: pacemakers, implanted medical pumps, metal plate in skull, metal objects inside the eye or skull, history of seizures.

Contraindications for MRI: pacemakers, brain stimulators, dental implants or metallic braces, aneurysm clips (metal clips on the wall of a large artery), metallic prostheses (including metal pins and rods, heart valves, and cochlear implants), permanent eyeliner, insulin pump, or shrapnel fragments. Welders and metal workers are also at risk for injury because of possible small metal fragments in the eye of which they may be unaware. Subjects will be screened for these contraindications prior to the study.

Subjects with previous or current neuropsychiatric disorders will be excluded. Patients with MRI findings consistent with organic brain lesions such as brain tumors, stroke, or trauma will be excluded. Patients with a history of significant medical disorders such as cancers will be excluded. Subjects not capable of giving informed consent will be excluded.

We will not scan pregnant women with MRI because safety of high magnetic field to fetus is not established. Therefore, we will administer a urine pregnancy test for any female subject of childbearing potential prior to MRI scan.

Brain functions at a development stage are out of scope of this particular experiment, and, therefore, subjects under age 21 will be excluded.

Subjects who show evidence of unusually increased cortical excitability that may lead to seizure activity detected by surface EMG recording will be excluded from the study. Subjects who always reveal muscle activity during the motor imagery task will also be excluded from the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20
Dates: Start 2002-09; Study Completion 2003-11

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Catalan MJ, Honda M, Weeks RA, Cohen LG, Hallett M. The functional neuroanatomy of simple and complex sequential finger movements: a PET study. Brain. 1998 Feb;121 ( Pt 2):253-64. doi: 10.1093/brain/121.2.253. PMID 9549504
- [Background] Cohen LG, Weeks RA, Sadato N, Celnik P, Ishii K, Hallett M. Period of susceptibility for cross-modal plasticity in the blind. Ann Neurol. 1999 Apr;45(4):451-60. doi: 10.1002/1531-8249(199904)45:43.0.co;2-b. PMID 10211469
- [Background] Classen J, Witte OW, Schlaug G, Seitz RJ, Holthausen H, Benecke R. Epileptic seizures triggered directly by focal transcranial magnetic stimulation. Electroencephalogr Clin Neurophysiol. 1995 Jan;94(1):19-25. doi: 10.1016/0013-4694(94)00249-k. PMID 7530636